CLINICAL TRIAL: NCT00689195
Title: Evaluation of Curcumin Formulation, and Ashwagandha Root Powder Extract in the Management of Advanced High Grade Osteosarcoma"
Brief Title: Pilot Study of Curcumin Formulation and Ashwagandha Extract in Advanced Osteosarcoma
Acronym: OSCAT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Pharmanza Herbals Pvt Limited (PHPL) (Unknown)
Responsible Party: Dr Manish Agarwal, Tata Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 381
Record Dates: First submitted 2008-05-23; First posted 2008-06-03 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Osteosarcoma
Keywords: Curcumin; Ashwagandha; osteosarcoma; Pharmacokinetics of curcumin and ashwagandha formulation; response
MeSH Terms: conditions — Osteosarcoma | interventions — Ashwagandha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C (Experimental): Curcumin
  Interventions: Dietary Supplement: Curcumin powder
- A (Experimental): Ashwagandha extract
  Interventions: Dietary Supplement: Ashwagandha extract

INTERVENTIONS:
Dietary Supplement: Curcumin powder — oral capsules containing the investigational agent
  Other Names: M3CX,
  Arms: C
Dietary Supplement: Ashwagandha extract — 4.5% extract of ashwagandha
  Other Names: Withania somnifera,; Dunal,; Indian Ginseng
  Arms: A

SUMMARY:
Curcumin as well as the ashwagandha extract are ingredients from traditional indian medicine and have been shown to be potent anti-cancer compounds in laboratory as well as animal studies. This study will test the safety and efficacy of a curcumin formulation and the ashwagandha extract in high grade relapsed or metastatic osteosarcoma where no other second line chemotherapy is being given. The pharmacokinetics will be studied along with response as measured on CT scans and PET scans as well as the quality of life and any toxicity.

DETAILED DESCRIPTION:
Eligibility criteria

1. Osteosarcoma which has relapsed after treatment and for which no second line chemotherapy is planned and in which disease is not amenable to surgery.
2. Patient should be able to follow-up 3 monthly for clinical and imaging assessment as well as biochemical tests

ELIGIBILITY:
Inclusion Criteria:

* Patients (between the ages of 8 to 65 years) with histologically proven high grade osteosarcoma of the extremity and relapsed disease after primary line of treatment who are unsuitable or refuse secondary chemotherapy.
* Patients with advanced disease unable or unwilling to take primary conventional treatment
* Patients with early or non-metastatic disease who are unable or unwilling to take the standard chemotherapy.
* Adequate hepatic function defined by total bilirubin not more than 1.5 times the upper limit of normal (ULN) and SGOT and SGPT not more than 2.5 times the (ULN)
* Adequate renal function defined by the creatinine clearance greater than 50 ml/min, calculated by cockcroft-Gault formula

Exclusion Criteria:

* Patients who are suitable for second line chemotherapy and can afford it
* Age less than 8 years or greater than 65 years
* Pregnant or lactating women
* Patients who are unable or unwilling to provide blood samples for the drug assays.
* Low grade osteosarcoma
* Patient requiring treatment with CYP3A4 inducers or inhibitors (patients on treatment for epilepsy or tuberculosis)
* Participation in any investigational drug study within 28 days prior to study treatment.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
response, toxicity, disease progression | 2 years

SECONDARY OUTCOMES:
quality of life | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India